CLINICAL TRIAL: NCT06442449
Title: Open-labeled, Randomized, Controlled Phase IV Clinical Trial to Evaluate the Immunogenicity and Safety of Booster Dose of sIPV Co-administered With MMR and HepA-I.
Brief Title: Booster Dose of sIPV Co-administered With MMR and HepA-I.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-sIPV-4003
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2024-05

CONDITIONS: Poliomyelitis
Keywords: sIPV; immunogenicity; safety; Combination Vaccination
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Trial group 1 (Experimental): vaccination with sIPV+MMR
  Interventions: Biological: sIPV; Biological: MMR
- Trial group 2 (Experimental): vaccination with sIPV+HepA-I
  Interventions: Biological: sIPV; Biological: HepA-I
- Control group 1 (Active Comparator): vaccination with sIPV
  Interventions: Biological: sIPV
- Control group 2 (Active Comparator): vaccination with MMR
  Interventions: Biological: MMR
- Control group 3 (Active Comparator): vaccination with HepA-I
  Interventions: Biological: HepA-I

INTERVENTIONS:
Biological: sIPV — vaccination with sIPV
  Arms: Control group 1; Trial group 1; Trial group 2
Biological: MMR — vaccination with MMR
  Arms: Control group 2; Trial group 1
Biological: HepA-I — vaccination with HepA-I
  Arms: Control group 3; Trial group 2

SUMMARY:
This is an Open-labeled, Randomized, Controlled Phase IV Clinical Trial to Evaluate the Immunogenicity and Safety of Booster Dose of Sabin Strain Inactivated Poliovirus Vaccine (Vero cell) (sIPV) Co-administered with Measles, Mumps, Rubella (MMR) Combined Live Attenuated Vaccine and Inactivated Hepatitis A (Hep-A) Vaccine.

DETAILED DESCRIPTION:
The trial plans to enroll 960 infants aged 18 months (+4 months) who had completed three primary doses of sIPV vaccine and were assigned in a 2:2:2:1:1 ratio to four groups including trial group 1, trial group 2, control group 1, control group 2, control group 2, with informed consent from the participant's guardian. Trial group 1 receive one dose of sIPV co-administered with one dose of MMR vaccine. Trial group 2 receive one dose of sIPV co-administered with one dose of inactivated hepatitis A vaccine. Control group 1 receive one dose of sIPV, control group 2 receive one dose of MMR vaccine, and control group 3 receive one dose of inactivated hepatitis A vaccine. About 3.0 ml of venous blood will be collected from all participants before and 30 days after vaccination for antibody detection. Immediate reactions will be observed for 30 minutes after vaccination, and adverse events occured from 0 to day 30 after vaccination will be collected.

ELIGIBILITY:
Inclusion Criteria:

* (1) healthy toddlers aged 18 months (+4 months);
* (2) completed three doses of sIPV primary immunization;
* (3) completed one dose of MMR vaccination;
* (4) able to provide proof of vaccination;
* (5) able to provide legal proof of identity;
* (6) The guardians of the participants were able to understand and agree to sign the informed consent.

Exclusion Criteria:

* (1) a history of vaccination with a polio-containing vaccine component in addition to three sIPV primary doses, according to the vaccination certificate;
* (2) have received a second dose of MMR vaccine or a vaccine containing a vaccine for measles, mumps or rubella, or hepatitis A vaccine (inactivated or attenuated), according to the vaccination certificate;
* (3) previous history of polio or measles or mumps or rubella or hepatitis A;
* (4) known severe allergy to the vaccine or vaccine components, such as urticaria, dyspnea, angioedema;
* (5) severe congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* (6) with autoimmune diseases or immunodeficiency diseases (including but not limited to systemic lupus erythematosus, asplenia, functional asplenia, and HIV infection);
* (7) abnormal coagulation function (such as coagulation factor deficiency, platelet abnormality), or obvious bleeding, hematoma, or ecchymosis after previous intramuscular injection or venipuncture;
* (8) have/have had a serious neurological disease (e.g., encephalopathy, epilepsy, convulsions [other than febrile convulsions]) or psychosis, a family history of neurological disease or psychosis;
* (9) receiving immunosuppressive or other immunomodulatory therapy, cytotoxic therapy within the past 6 months, or planning to receive such treatment during the trial;
* (10) have received an immune globulin or other blood products within the past 6 months or plan to receive such treatment during the trial;
* (11) receipt of other investigational vaccines within 30 days before vaccination with the investigational vaccines;
* (12) receipt of live attenuated vaccine within 28 days before vaccination with the investigational vaccine;
* (13) receipt of subunit or inactivated vaccine within 7 days before vaccination with the investigational vaccine;
* (14) acute diseases or acute episodes of chronic diseases within the past 7 days;
* (15) Axillary temperature >37.0℃ if fever occurred before vaccination;
* (16) which are unsuitable for participation in the clinical trial as judged by the investigators.

Ages: 18 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 889 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
seroconversion rates (SCRs) of sIPV neutralizing antibody against different poliovirus serotypes (Type I, II and III) | 30 days
  -The SCRs of neutralizing antibody against different poliovirus serotypes (Type I, II and III) at day 30 after sIPV vaccination.
SCRs of anti-meascles IgG antibodies | 30 days
  SCRs of anti-measles IgG antibodies 30 days after vaccination
SCRs of anti-mumps IgG antibodies | 30 days
  SCRs of anti-mumps IgG antibodies 30 days after vaccination
SCRs of anti-rubella IgG antibodies | 30 days
  SCRs of anti-rubella IgG antibodies 30 days after vaccination
SCRs of anti-hepatitis A IgG antibodies | 30 days
  SCRs of anti-hepatitis A antibodies 30 days after vaccination

SECONDARY OUTCOMES:
Seropositivity rates (SPRs) and GMC of anti-measles virus IgG antibodies | 30 days
  SPRs and GMC of anti-measles virus IgG antibodies 30 days after vaccination.
SPRs and GMC of anti-mumps virus IgG antibodies | 30 days
  SPRs and GMC of anti-mumps virus IgG antibodies 30 days after vaccination;
SPRs and GMC of anti-rubella virus IgG antibodies | 30 days
  SPRs and GMC of anti-rubella virus IgG antibodies 30 days after vaccination;
SPRs and GMC of anti- hepatitis A virus IgG antibodies | 30 days
  SPRs and GMC of anti- hepatitis A virus IgG antibodies 30 days after vaccination;
Geometric Mean Titer (GMT) of sIPV neutralizing antibody against different poliovirus serotypes (Type I, II and III) | 30 days
  -GMTs of antibody of neutralizing antibody against different poliovirus serotypes (Type I, II and III) at day 30 after sIPV vaccination;
- SPRs of neutralizing antibodies against different poliovirus serotypes (Type I, II and III) | 30 days
  - SPRs of neutralizing antibodies against different poliovirus serotypes (Type I, II and III) at day 30 after vaccination.
- Incidence of adverse reactions (ARs) | 30 days
  - Incidence of ARs from 0 to 30 days after vaccination;
- Incidence of serious adverse events (SAEs) | 30 days
  - Incidence of SAEs 0~30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Pan Hongxing, Principal Investigator — Jiangsu Center for Disease Control and Prevention (Jiangsu Institute of Public Health)
Locations (1):
- Jiangsu Center for Disease Control and Prevention (Jiangsu Institute of Public Health), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu J, Han W, Chu K, Zhang H, Tuo L, Duan X, Li J, Yuan F, Luan C, Pan H, Jiao P. Immunogenicity and Safety of Sabin Strain Inactivated Poliovirus Vaccine Booster Dose Administered Separately or Concomitantly with Inactivated Hepatitis A Vaccine or Measles-Mumps-Rubella Combined Attenuated Live Vaccine: An Open-Labelled, Randomized, Controlled, Phase 4 Clinical Trial. Vaccines (Basel). 2025 Oct 23;13(11):1087. doi: 10.3390/vaccines13111087. PMID 41295459